CLINICAL TRIAL: NCT05176210
Title: A Phase I, Double-Blind, Placebo-Controlled, Randomized, Single- and Multiple-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Food Effect and Potential Efficacy of PS1 in Subjects
Brief Title: Safety, Pharmacokinetics, and Food Effect of PS1 in Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmasaga Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: PS1-01
Record Dates: First submitted 2021-11-29; First posted 2022-01-04 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Type II Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 5-tert-butyl-N-pyrazol-4-yl-4,5,6,7-tetrahydrobenzo(d)isoxazole-3-carboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- SAD portion - Cohort 1 (25mg) (Experimental): An eligible subject will receive a single dose of 25 mg of PS1 or Placebo tablets in a fed condition on Day 1 and be followed for 7 days.
  Interventions: Drug: PS1; Drug: Placebo
- SAD portion - Cohort 2 (50mg) (Experimental): An eligible subject will receive a single dose of 50 mg of PS1 or Placebo tablets in a fed condition on Day 1 and be followed for 7 days.
  Interventions: Drug: PS1; Drug: Placebo
- SAD portion - Cohort 3 (75mg) (Experimental): An eligible subject will receive a single dose of 75 mg of PS1 or Placebo tablets in a fed condition on Day 1 and be followed for 7 days.
  Interventions: Drug: PS1; Drug: Placebo
- FE portion - Cohort 4 (50mg) (Experimental): An eligible subject will receive a single dose of 50 mg PS1 or Placebo tablets in a fasted condition on Day 1 and be followed for 7 days.
  Interventions: Drug: PS1; Drug: Placebo
- MAD portion - Cohort 5 (25mg) (Experimental): An eligible subject will receive 25 mg PS1 or Placebo tablets once daily in a fed condition for 14 days and be followed for additional 7 days.
  Interventions: Drug: PS1; Drug: Placebo
- MAD portion - Cohort 6 (50mg) (Experimental): An eligible subject will receive 50 mg PS1 or Placebo tablets once daily in a fed condition for 14 days and be followed for additional 7 days.
  Interventions: Drug: PS1; Drug: Placebo
- MAD portion - Cohort 7 (25mg) (Experimental): An eligible subject will receive 25 mg PS1 or Placebo tablets once daily in a fed condition for 28 days and be followed for additional 7 days.
  Interventions: Drug: PS1; Drug: Placebo
- MAD portion - Cohort 8 (50mg) (Experimental): An eligible subject will receive 50 mg PS1 or Placebo tablets once daily in a fed condition for 28 days and be followed for additional 7 days.
  Interventions: Drug: PS1; Drug: Placebo

INTERVENTIONS:
Drug: PS1 — PS1 will be provided as a 120 mg tablet with 25 mg active pharmaceutical ingredient.
  Other Names: PS-001
Drug: Placebo — Placebo will be provided as a 120 mg tablet.

SUMMARY:
This is a phase I, double-blind, placebo-controlled, randomized, single- and multiple-ascending dose study to evaluate new study intervention, PS1. PS1 is a potential blood glucose control medication, which is developed by Pharmasaga Co. Ltd. planned for treating type II diabetes mellitus (T2DM). This is a first-in-human study to evaluate the safety, tolerability, pharmacokinetics (PK), food effect and potential efficacy of PS1 in subjects.

DETAILED DESCRIPTION:
This first-in-human Phase I study consists of a single ascending-dose (SAD) portion, a food effect (FE) portion, and a multiple ascending-dose (MAD) portion, aiming to evaluate the safety, tolerability, pharmacokinetics, food effect and potential efficacy of PS1 in healthy subjects.

A randomized, double-blinded, placebo-controlled study design will be applied for the SAD portion with three SAD dose cohorts-25 mg (Cohort 1), 50 mg (Cohort 2), and 75 mg (Cohort 3). An eligible subject in this portion will receive a single dose of PS1 or Placebo tablets in a fed condition on Day 1 and be followed for 7 days.

In FE portion, only one cohort (Cohort 4) is assigned. The FE cohort (Cohort 4) will use the same study design as the SAD cohorts. An eligible subject in this portion will receive a single dose of 50 mg PS1 or Placebo tablets in a fasted condition on Day 1 and be followed for 7 days.

Four cohorts are assigned in the MAD portion: 25 mg/day (Cohort 5 & 7) and 50 mg/day (Cohort 6 & 8) in healthy volunteers and participants respectively. Only the dose level of MAD lower than the maximum tolerated dose (MTD) of SAD portion can be activated (If 50 mg was determined as the MTD of SAD, only cohort 5 & 7 could be activated). An eligible subject will receive PS1 or Placebo tablets once daily in a fed condition for 14 days & 28 days in healthy volunteers and participants respectively and be followed for additional 7 days.

ELIGIBILITY:
Inclusion Criteria:

For all cohorts, a subject is eligible for the study if all of the following apply:

1. Both genders aged 18 to 80 years, inclusive at screening
2. Body mass index (BMI) between 18.5 and 40.0 kg/m2
3. Negative test for hepatitis B surface antigen (HBsAg), Anti-HCV antibody, and human immunodeficiency virus (HIV) at screening
4. Is willing to follow the trial life style instruction and protocol procedure
5. Able to understand and sign the informed consent form.

   Inclusion criteria applied for healthy subjects (Cohorts 1~6)
6. Overtly healthy subject, who is considered to be generally healthy based on medical history, vital signs, laboratory tests, 12-lead EKG, and physical examination, as judged by the investigator
7. With HbA1c value of < 6.5% and fasting plasma glucose < 110 mg/dL at Screening
8. With estimated glomerular filtration rate (eGFR) > 80 ml/min

   Inclusion criteria applied for T2DM patients (Cohort 7 and 8)
9. Diagnosis of T2DM
10. T2DM treated with diet and exercise alone currently, for at least 2 weeks prior to Screening
11. With HbA1c level between 6.5% to 9.0% and fasting plasma glucose level between 130 mg/dL to 250 mg/dL at Screening
12. With estimated glomerular filtration rate (eGFR) > 60 ml/min
13. For patients taking medication for other chronic disease, the medication should be on a stable dose for at least 4 weeks prior to Screening, and should not be a strong CYP enzyme inhibitor or inducer

Exclusion Criteria:

For all cohorts, a subject meeting any of the following exclusion criteria will be excluded from study participation.

1. History of Type I diabetes mellitus
2. Under the systemic treatment of any prescription medication or over-the-counter (OTC) medication that may interfere with the safety or PK assessment judged by the investigator within 7 days before Screening
3. Received strong CYP enzyme inhibitor or inducer within 14 days before Screening
4. Received any vaccination within 14 days before Screening
5. Has required insulin therapy within the past 12 weeks
6. Known hypersensitivity to any of the components of PS1 tablet
7. History of major clinically significant hematological, renal, respiratory, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, musculoskeletal, immune, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing) within 3 months of Screening that may significantly alter the biomarker panel, require receiving any systemic medications, or interfere with the interpretation of data, as judged by the investigator
8. History of pancreatitis
9. Serum amylase > 1.5 × Upper Limit of Normal (ULN) or lipase > 1.5 × ULN
10. Clinically significant ECG abnormality at Screening
11. History of cancer (malignancy) or have ever received any anti-cancer therapy
12. Regular smoker Regular smoker is defined as who smokes every day (≥ 1 cigarette/day in average in the past 8 weeks of Screening)
13. Consumed greater than 3 units of alcoholic beverages per day in average for the past 4 weeks before Screening One unit is equivalent to one can of beer (20% alcohol; about 45 mL)
14. Received any investigational therapy from another clinical study or underwent any major surgeries within the last 12 weeks prior to Screening.
15. Took glucose-lowering medications within the last 2 weeks prior to Screening
16. Received any systemic steroids (inhaled and intranasal steroids are permitted) or other immunosuppressive medications within 4 weeks prior to Screening
17. Have ever received cell therapy or organ transplantation
18. Other conditions not suitable for participating in this study as judged by the investigator
19. Any conditions that forbid the completion of study procedures due to the local regulatory restrictions
20. Female subject of childbearing potential who:

    * Is lactating; or
    * Has a positive pregnancy test result at Screening; or
    * Refuses to adopt at least one form of birth control (refer to Section 5.3) from signing informed consent to the end of the study.
21. Male subject with a female spouse/partner who is of childbearing potential refuses to adopt at least one form of birth control (refer to Section 5.3) from signing informed consent to the end of the study.

    Exclusion criteria applied for healthy subjects (Cohorts 1~6):
22. History of type II diabetes mellitus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-12-22 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) during the DLT observation period | Day 1~ Day 8 (SAD cohort); Day 1~ Day 35 (MAD cohort)
  DLT is defined as: (1) any adverse event (AE) ≥ Grade 3 (CTCAE v5.0) or (2) Grade 2 AE that does not resolve to grade 1 or less within 72 hours, that occurs in the DLT observation period and is causally related (possibly, probably, or definitely related) to the test article judged by the investigator.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) | SAD, FE: up to 4 weeks; MAD: up to 8 weeks
  All adverse events (AEs) will be assessed for severity by the investigator based on NCI-CTCAE v5.0
Number of participants with abnormalities in Vital signs | SAD, FE: Baseline,1~2 weeks; MAD: Baseline,1~6 weeks
  Number of participants with abnormal systolic/diastolic blood pressure (in mmHg), respiratory rate, pulse rate (in beat per minute, bpm), and body temperature (in ℃)
Number of participants with abnormalities in Laboratory examinations | SAD, FE: Baseline,1~2 weeks; MAD: Baseline,1~6 weeks
  Number of participants with abnormal Hematology (hemoglobin, hematocrit, RBC, platelet, WBC, WBC differentials (neutrophils, eosinophils, basophils, lymphocytes, monocytes), MCV, MCH, MCHC), biochemistry (HbA1c, fasting plasma glucose, albumin, alkaline phosphatase, ALT, AST, BUN, creatinine, cholestero1, γ-GT, total protein, total bilirubin, direct bilirubin, triglyceride, amylase, lipase, calcium, sodium, potassium, chloride), and urinalysis (pH, protein, glucose, bilirubin, urobilinogen, ketone body, specific gravity, occult blood, RBC, WBC, creatinine, ratio of albumin/creatinine) results
Acute kidney injury (AKI) marker | SAD, FE: Baseline, 1~2 weeks; MAD: Baseline, 1~6 weeks
  Urine samples will be collected for analyzing acute kidney injury (AKI) markers
Number of participants with abnormalities in 12-lead electrocardiogram (EKG) | SAD, FE: Baseline, 1~2 weeks; MAD: Baseline, 1~6 weeks
  Number of participants with abnormal Ventricular rate, PR interval, QRS interval, and QT interval
Number of participants with abnormalities in Physical examination | SAD, FE: Baseline, 1~2 weeks; MAD: Baseline, 1~6 weeks
  Number of participants with abnormal Physical examination results, including general appearance, skin, eyes, ears, nose, throat, head and neck (including thyroid), heart, chest and lungs, abdomen, extremities, lymph nodes, musculoskeletal, neurological system, and other body systems
Pharmacokinetics (PK) of PS1 | Day 1 and 2 (SAD, FE and MAD portion), Day 28 and 29 (MAD portion only)
  AUC_Area under the serum concentration-time profile
Pharmacokinetics (PK) of PS1 | Day 1 and 2 (SAD, FE and MAD portion), Day 28 and 29 (MAD portion only)
  Cmax_The peak post-dose concentration
Pharmacokinetics (PK) of PS1 | Day 1 and 2 (SAD, FE and MAD portion), Day 28 and 29 (MAD portion only)
  Tmax_Time at which Cmax is observed
Pharmacokinetics (PK) of PS1 | Day 1 and 2 (SAD, FE and MAD portion), Day 28 and 29 (MAD portion only)
  T1/2_Terminal phase elimination half-life
Pharmacokinetics (PK) of PS1 | Day 1 and 2 (SAD, FE and MAD portion), Day 28 and 29 (MAD portion only)
  MRT_Mean Residence Time
Pharmacokinetics (PK) of PS1 | Day 1 and 2 (SAD, FE and MAD portion), Day 28 and 29 (MAD portion only)
  CL/F_Apparent Clearance
Pharmacokinetics (PK) of PS1 | Day 1 and 2 (SAD, FE and MAD portion), Day 28 and 29 (MAD portion only)
  Volume of distribution
Pharmacokinetics (PK) of PS1 | Day 1 and 2 (SAD, FE and MAD portion), Day 28 and 29 (MAD portion only)
  Rac_Accumulation ratio
Potential efficacy (For Cohort 7 and 8 only) | MAD: Baseline, 1~6 weeks
  Changes from baseline of fasting plasma glucose (FPG) at each post-treatment visit; Changes from baseline of C-peptide at each post-treatment visit; Changes from baseline of hemoglobin A1c (HbA1c) at Visit 10 and Visit 11.
Exploratory Endpoints (For MAD only) | MAD: Baseline, 1~6 weeks
  Changes from baseline of serum PDIA4

CONTACTS AND LOCATIONS:
Overall Officials: Mingche Liu, MD., PhD, Principal Investigator — Taipei Medical University Hospital
Locations (1):
- Mingche Liu, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No